CLINICAL TRIAL: NCT06860542
Title: Inhaled Budesonide for REcurrence Prevention and Adjuvant THerapy in Checkpoint Inhibitor Pneumonitis
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: AHS Cancer Control Alberta (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IBREATHCIP
Record Dates: First submitted 2025-02-24; First posted 2025-03-06 (Actual); Last update posted 2025-09-25 (Actual); Status verified 2025-09

CONDITIONS: Pneumonitis; Immune-related Adverse Event
Keywords: Immune-related Adverse Event; Checkpoint Inhibitor Pneumonitis
MeSH Terms: conditions — Pneumonia

STUDY DESIGN:
Intervention Model Description: Budesonide (Pulmicort® Turbuhaler®) 800ug inhaled twice daily (BID) will be taken in addition to usual care for 36 weeks. Checkpoint inhibitor pneumonitis (CIP) flare/recurrence will be treated as initial episode/per guidelines.
  The comparison arm will be usual care (UC) for CIP; recommended guideline management consists of systemic steroids 1-2mg/kg via oral (grade 2) or intravenous (IV) (grade 3/4) until clinical improvement, then taper over 6 weeks (grade 2) or 8 weeks (grade 3/4). Final CIP management decisions at treating physicians discretion.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Arm 1- Usual care (Active Comparator): The comparison arm will be usual care (UC) for Checkpoint Inhibitor Pneumonitis (CIP); recommended guideline management consists of systemic steroids 1-2mg/kg via oral (grade 2) or IV (grade 3/4) until clinical improvement, then taper over 6 weeks (grade 2) or 8 weeks (grade 3/4). Final CIP management decisions at treating physicians discretion.
  Interventions: Other: Arm 1- Usual care
- Arm 2- Budesonide (Pulmicort® Turbuhaler®) + Usual care (Experimental): Budesonide (Pulmicort® Turbuhaler®) 800ug inhaled twice daily (BID) will be taken in addition to usual care for 36 weeks. Checkpoint Inhibitor Pneumonitis (CIP) flare/recurrence will be treated as initial episode/per guidelines.
  Interventions: Drug: Arm 2- Budesonide (Pulmicort® Turbuhaler®) + Usual care

INTERVENTIONS:
Drug: Arm 2- Budesonide (Pulmicort® Turbuhaler®) + Usual care — Budesonide (Pulmicort® Turbuhaler®) 800ug inhaled twice daily (BID) will be taken in addition to usual care for 36 weeks.
  Arms: Arm 2- Budesonide (Pulmicort® Turbuhaler®) + Usual care
Other: Arm 1- Usual care — The comparison arm will be usual care (UC) for Checkpoint inhibitor pneumonitis (CIP) (steroids).
  Other Names: Comparator arm
  Arms: Arm 1- Usual care

SUMMARY:
The introduction of immune checkpoint inhibitors (immunotherapy) that stimulate our immune system to recognize and attack cancer cells has been one of the most exciting advances in oncology over the last decade. These medications are now employed across almost half of cancer types and settings, however they come with a cost. In some patients, instead of attacking cancer cells alone, the stimulated immune system damages healthy tissues (immune related adverse events), with one of the most severe and potentially deadly such complications being immune attack on the lungs, or checkpoint inhibitor pneumonitis (CIP). When treated promptly with oral or intravenous steroids, acute CIP improves in many cases, however for approximately one-fifth of patients the lung inflammation is difficult to control, resulting in recurrent shortness of breath, the need for extended courses of oral or intravenous steroids, impacting quality of life and cancer therapy decisions. The goal of the trial is to assess whether use of inhaled steroids, a type of medication commonly used in asthma patients, for one year after a first diagnosis of CIP may help the lung inflammation resolve and not return, without the repeated use of oral or intravenous medications that carry more side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients must be 18 years of age, or older on the day of signing informed consent and be willing and able to provide written informed consent/assent and, in the opinion of the Investigator, comply with protocol tests and procedures
2. Patients require histologically confirmed solid tumour undergoing immune checkpoint inhibitor (ICI) therapy
3. Diagnosis of first documented diagnosis of Checkpoint Inhibitor Pneumonitis (CIP) made per European Society for Medical Oncology (ESMO)/American Society for Medical Oncology (ASCO) guidelines with severity >/grade 2 by Common Terminology Criteria for Adverse Events (CTCAE)v5.0

   a. Per ASCO/ESMO consensus guidelines, workup must include a compatible clinical picture, plus/minus supporting radiographic evidence (chest x-ray or preferably computed tomography (CT)), combined with clinical and/or microbiologic ruling out of alternative etiologies including infections or pulmonary disease progression. This includes a negative COVID test. Bronchoscopic sampling is not required, but can be considered.
4. Be able to effectively operate and use budesonide delivery method (Turbuhaler®), either independently or with aid of caregiver who anticipates being able to do so throughout trial period
5. Have adequate organ function, as judged by enrolling clinician
6. Females of childbearing potential have a negative urine or serum pregnancy test prior to study day 1. Patients of childbearing potential are those who have not been surgically sterilized or have not been free of menses for at least 1 year
7. Females of childbearing potential are willing to use contraception or abstain from heterosexual sexual contact for the course of the study

Exclusion Criteria:

1. Diagnosis of interstitial lung disease (ILD) active (clinically and radiologically evident) within last year prior to diagnosis of CIP
2. Clinically suspected significant lung disease for which inhaled steroid would be standard of care (moderate asthma or severe chronic obstructive pulmonary disease (COPD)) and for which randomization to no inhaled steroids (control arm) would not represent optimal medical care. Based on enrolling physicians judgement; spirometry/pulmonary function tests are NOT required to assess this exclusion criteria.
3. Current (within last two weeks), active (not medically able or unwilling to discontinue prior to treatment start) and regular (2 or more times per week) use of inhaled steroids (for any indication) or systemic (>10mg prednisone equivalent) corticosteroids (for indication other than CIP) at time of randomization
4. Receiving systemic, non-chemotherapy immunosuppressive agent at time of randomization (hydroxychloroquine is acceptable)
5. Use of a medication with significant interaction with inhaled budesonide (HIV protease inhibitors, ketoconazole or other potent CYP3A4 inhibitors), unless deemed required and safe by co-investigator.
6. Known poorly controlled diabetes, defined as A1c >10, prior to initiation of steroids for CIP
7. History of active and unstable systemic disease, including heart failure New York Heart Association (NYHA) III or IV, cirrhosis with Child Pugh B or C, Renal Failure with creatinine clearance (CrCl) <30 per Cockcroft-Gault formula, or other unstable life limiting condition as determined by trial investigators
8. Current or prior participation in a study of an investigational agent or device within 4 weeks of randomization
9. History or current evidence of any condition, therapy, or laboratory abnormalities which might confound trial results, interfere with the patient's participation for the full duration of the trial, or otherwise causing it to be not in the best interest of the patient to participate in the trial, in the opinion of the treating investigator.
10. Is or has an immediate family member (e.g., spouse, parent/legal guardian, sibling or child) who is directly involved with this trial, unless prospective ethics board approval (by chair or designee) is given allowing exception to this criterion for a specific patient
11. Breastfeeding is not permitted during the duration of trial participation.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 94 (Estimated)
Dates: Start 2025-12-01 (Estimated); Primary Completion 2029-12-01 (Estimated); Study Completion 2030-12-01 (Estimated)

PRIMARY OUTCOMES:
Assess efficacy of inhaled budesonide in reducing the development of refractory or recurrent Checkpoint Inhibitor Pneumonitis (RR-CIP) after initial episode of >/grade 2 CIP | 1 year
  Compare incidence of refractory or recurrent Checkpoint inhibitor pneumonitis (RR-CIP) after initial episode of >/grade 2 CIP with or without addition of inhaled budesonide to usual care.

SECONDARY OUTCOMES:
Assess steroid toxicities after development of >/grade 2 Checkpoint inhibitor pneumonitis (CIP) | 1 year
  Frequency of grade 2 or higher steroid toxicities (systemic and local for inhaled) by 36 weeks with or without inhaled budesonide in addition to standard of care in patients after development of >/grade 2 CIP. Safety of intervention will be assessed with this endpoint, but importantly this will also assess any reduction of systemic steroid side effects
Compare systemic steroids requirements in patients after development of >/grade 2 Checkpoint inhibitor pneumonitis (CIP) | 1 year
  Total dose of systemic steroids (mg/kg prednisone equivalents) required by patients at 36 weeks with or without inhaled budesonide after development of >/grade 2 CIP (interim analysis planned). Total dose calculated from start of first systemic steroid taper.
Assess the impact of adjuvant inhaled budesonide on time to improvement of initial episode of Checkpoint inhibitor pneumonitis (CIP) | 1 year
  Time to symptomatic improvement after initial episode of CIP with or without inhaled budesonide, as assessed by time to improvement by Modified Medical Research Council (mMRC) dyspnea level(s) and Common Terminology Criteria for Adverse Events (CTCAE) v5.0 pneumonitis grade(s).
Compare Patient Reported Outcomes (PROs) in patients after initial episode of Checkpoint inhibitor pneumonitis (CIP) | 1 year
  Trends of Patient Reported Outcomes (PROs) with or without inhaled budesonide assessed by Patient-Reported Outcomes Version of the Common Terminology Criteria for Adverse Events (PRO-CTCAE) v1.0 at 8 week intervals

IPD SHARING:
Plan to Share IPD: No